CLINICAL TRIAL: NCT07277543
Title: Assessment of Dentoskeletal Changes After Treatment of Skeletal classII Growing Patient by Twinblock Versus Monoblock Appliance
Brief Title: Assessment of Dentoskeletal Changes After Treatment of Skeletal classII by Twinblock Versus Monoblock Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Shimaa Nasr, principle investigator, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-108-2-H
Record Dates: First submitted 2025-11-16; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Dentoskeletal Changes in Skeletal classII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment of skeletal classII by twin block (Experimental): growing patient wearing twin block appliance15 hrs/day
  Interventions: Device: wearing of twinblock after bite correction
- treatment of skeletal classII by monoblock (Experimental): growing patients wearing monoblck appliance15hrs/day
  Interventions: Device: wearing of monoblock after bite correction

INTERVENTIONS:
Device: wearing of twinblock after bite correction — bite registration at edge to edge position ,twin block wearing 15hrs/day
  Arms: treatment of skeletal classII by twin block
Device: wearing of monoblock after bite correction — bite registration at edge to edge position ,mono block wearing 15hrs/day
  Arms: treatment of skeletal classII by monoblock

SUMMARY:
Assessment of dentoskeletal changes after treatment of skeletal classII growing patient by twin block versus mono block ,clinical trial stuy

DETAILED DESCRIPTION:
Group(A):patients will be treated with twinbLock Group(B):patients will be treated with monobLock

ELIGIBILITY:
Inclusion Criteria:

* Female patients to avoid any sexual dimorphism which may affect the comparison.
* Skeletal Class II (ANB° > 5°) with normal maxilla (SNA° = 82° ±4°) and retrognathic mandible (SNB° < 87°).
* Age range from 9 to 12 years.

Exclusion Criteria:

* Previous history of orthodontic treatment.
* Congenitally missing or extracted permanent teeth.
* Posterior cross bites or severe maxillary transverse deficiency.
* Severe facial asymmetry determined by clinical or radiographic examination.
* Poor oral hygiene.
* Systemic diseases that may affect the treatment results.

Ages: 9 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
skeletal classII correction and dental changes | 8_12 month
  standerized extraoral radiograph and Cone-Beam Computed Tomography(CBCT)

SECONDARY OUTCOMES:
Assessment of airway changes | 8-12month
  cone beam computed tomography(cbct)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Mostafa Mohammed, Ass.Professor, Principal Investigator — Ass.Professor of Orthodontics
Locations (1):
- Shimaa Nasr, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sakuno AC, da Rosa APB, Maeda FA, Trivino T, Carvalho PEG, Torres FC. Tomographic evaluation of dentoskeletal changes due to the treatment of class II malocclusion with Forsus appliance. J Oral Biol Craniofac Res. 2019 Jul-Sep;9(3):277-279. doi: 10.1016/j.jobcr.2019.06.005. Epub 2019 Jun 5. PMID 31289716
- See also: evaluation of dentoskeletal changes due to the treatment of class II malocclusion — https://pubmed.ncbi.nlm.nih.gov/31289716/